CLINICAL TRIAL: NCT00364767
Title: The Effect of Moderate Alcohol Consumption on Markers of Oxidative Phosphorylation and Lipid Oxidation and on Postprandial Glycemic Control in Healthy, Lean and Overweight, Young Men
Brief Title: Moderate Alcohol Consumption, Fat and Carbohydrate Metabolism and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Collaborators: Dutch Foundation for alcohol research (Unknown)
Responsible Party: Henk Hendriks, TNO Quality of Life
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P5805
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Disease
Keywords: Moderate alcohol consumption; Fat and carbohydrate oxidative capacity; Postprandial glycemic response
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Whiskey (32 gram of alcohol/day)
  Interventions: Dietary Supplement: A
- B (Placebo Comparator): Water (0 gram alcohol/day)
  Interventions: Dietary Supplement: B

INTERVENTIONS:
Dietary Supplement: A — Alcohol consumption (32 g/day) for 4 weeks
  Arms: A
Dietary Supplement: B — Water
  Arms: B

SUMMARY:
Moderate alcohol consumption is associated with a decreased risk of diabetes type 2. This association could be mediated by an improvement of insulin sensitivity with moderate alcohol consumption. Patients with diabetes type 2 or impaired glucose tolerance often may have decreased fat oxidative capacity or oxidative phosphorylation in tissue such as muscle. This could lead to accumulation triglyceride storage in muscle, which could interfere with insulin signaling. Whether such mechanism can also play a role with moderate alcohol consumption is unknown and will be investigated in this study.

In addition, moderate alcohol consumption with a meal can lead to delayed hypoglycemia in type 1 diabetes patients. How moderate alcohol consumption affects postprandial glycemic response in healthy subjects is unknown. This is a secondary objective of this trial.

DETAILED DESCRIPTION:
To investigate the effect of moderate alcohol consumption on

* enzymes involved in fatty acid oxidation, oxidative phosphorylation and glycolysis in skeletal muscle
* transporters of fatty acids and glucose in fat tissue
* post-prandial glycemic response in healthy, lean or overweight, young men

Design : Open, randomized, partially diet-controlled, placebo controlled cross-over design

Participants

* Description : Healthy, lean and overweight young (18-40 years) men
* Number : 20

Study substances

* Test substance : 100 ml whiskey (Famous Grouse, 40% v/v alcohol: ≈ 32 g alcohol)
* Reference substance : 100 ml mineral water (Spa blauw)

Duration: 2 treatment periods of 4 weeks (28 days)

Test parameters:

* Muscle biopsy for activity of 3-hydroxy fatty-acyl CoA dehydrogenase, citrate synthase, cytochrome c oxidase
* Postprandial glycemic response (glucose, insulin, GLP-1, GLP-2, GIP, glucagon, FFA etc.)
* Insulin sensitivity and related factors (oral glucose tolerance test, adiponectin, HbA1c)
* Liver enzymes (safety)
* Body weight
* Urinary ethyl glucuronide (compliance)

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged between 18 and 40 years
* Lean subjects BMI 18.5-25 kg/m2 and overweight/obese subjects BMI >27 kg/m2 (including 18.5, 25 and 27)
* Alcohol consumption between 7 and 28 units/week (including 7 and 28)

Exclusion Criteria:

* Smoking
* Family history of alcoholism
* History of medical or surgical events that may significantly affect the study outcome, particularly metabolic or endocrine disorders and gastrointestinal disorders
* Recent blood donation
* More than 8 hours/week of intense exercise
* Blood haemoglobin concentration below 8.4 mmol/l
* Allergic to betadine or lidocaine.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
enzymes involved in fatty acid oxidation, oxidative phosphorylation and glycolysis in skeletal muscle | 4 weeks

SECONDARY OUTCOMES:
Post-prandial glycemic response | 4 weeks
insulin sensitivity (oral glucose tolerance test) and related factors (adiponectin, HbA1c) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Henk FJ Hendriks, PhD., Principal Investigator — TNO

REFERENCES:
- [Result] Beulens JW, van Loon LJ, Kok FJ, Pelsers M, Bobbert T, Spranger J, Helander A, Hendriks HF. The effect of moderate alcohol consumption on adiponectin oligomers and muscle oxidative capacity: a human intervention study. Diabetologia. 2007 Jul;50(7):1388-92. doi: 10.1007/s00125-007-0699-8. Epub 2007 May 11. PMID 17492425